CLINICAL TRIAL: NCT06711315
Title: Oral Mucositis Management Supported by MASCC/ISOO Protocols: A Randomized Controlled Trial in Pediatric Oncology Patients
Brief Title: Oral Mucositis Management in Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zubeyde Ezgi Ercelik (Other)
Responsible Party: Sponsor-Investigator, Zubeyde Ezgi Ercelik, Assistant Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023 - 695; From Researcher (Other: Bandırma Onyedi Eylül University)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Childhood Oncology; Mucositis Oral
Keywords: Childhood, cancer, oral mucosit, oral care
MeSH Terms: conditions — Stomatitis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Oral mucositis education was given, oral care was requested for 14 days and monitored on days 0, 3, 7 and 14.
  Interventions: Behavioral: Oral Mucosit Care Protocol
- Control Group (No Intervention): Children in the control group will receive standard care. Mouthwash with sodium bicarbonate (after each feeding), mycostatin (2x1) and tranflex (3x1). Toothbrush and dental floss are not used. At the end of the 14th day, the child and caregiver in the control group will receive Oral Care Protocol Training to Prevent Oral Mucositis.

INTERVENTIONS:
Behavioral: Oral Mucosit Care Protocol — The children in the intervention group were subjected to a four-stage intervention carried out by the nurse researcher. The practices in each stage were as follows.
  Stage 1: Oral care protocol training to prevent oral mucositis Stage 2: Introduction and application of training material (brochure) Stage 3: Introduction and implementation of oral care calendar Stage 4: Implementation of oral care protocol
  Arms: Intervention Group

SUMMARY:
This study evaluated the impact of an oral mucositis care protocol on the severity of mucositis.

The main questions it aims to answer are:

-What is the severity of mucositis in parents and children who receive oral mucositis education?

The data were collected using a descriptive information form, the Children's International Mucositis Evaluation Scale (ChIMES), and the WHO Oral Mucositis Grading Scale. Standard care was applied to the control group. For the intervention group, an oral care protocol was prepared, and the patients received training. The oral care intervention was applied for 14 days and monitored by the researcher. The patients were monitored for oral mucositis on Days 0, 3, 7, and 14. Those in the intervention group received a calendar for documenting their oral care practices.

DETAILED DESCRIPTION:
Data Collection Process The researchers informed children and their parents about the purpose of the study. Written and verbal consent was obtained from both willing children and their parents.

The researcher works as a nurse in the pediatric oncology clinic. If the children met the inclusion criteria, the researchers visited the clinics, introduced themselves to the child and the family, and provided information about the research. The child and the family were informed about the research. All caregivers (both intervention and control groups) who meet the inclusion criteria and agree to participate in the study will be asked to fill out the Descriptive Characteristics Form. Research data will be obtained by conducting four assessment interviews with each child and caregiver. The first interview will be conducted before the treatment, the second interview will be conducted on the 3rd day after the treatment, and the following interviews will be conducted on the 7th and 14th days of the treatment and the oral mucosa will be evaluated by the researcher by interviewing the child and caregiver and using scales.

The child and caregiver in the intervention group will receive an oral care protocol on days 0-14 of treatment. The child and caregiver in the control group will receive standard care.

Procedures Intervention Group The children in the intervention group were subjected to a four-stage intervention carried out by the nurse researcher. The practices in each stage were as follows.

Stage 1: Oral care protocol training to prevent oral mucositis Stage 2: Introduction and application of training material (brochure) Stage 3: Introduction and implementation of oral care calendar Stage 4: Implementation of oral care protocol

Stage 1: Oral care protocol training to prevent oral mucositis Oral care protocol was prepared according to the protocols to standardize oral care practices for children and caregivers before chemotherapy treatment. Expert opinions were collected to inform the content of the training, which was administered in a single session. The training session included a PowerPoint presentation identifying the definition of oral mucositis, the cause of occurrence, signs and symptoms, and the oral care protocol. Together with each child and their caregiver who completed the training, the researcher applied the oral care protocol and answered questions. All material to be applied in the oral care protocol. was introduced to each patient in a one-on-one meeting. At the end of the training, the participants received a training brochure containing the material and application steps. Separate trainings were given to each child hospitalized in the clinic and their caregiver.

Stage 2: Introduction and application of training material (brochure) The children received a brochure with directions for using the medicine and information about how many times it should be used per day.

Stage 3: Introduction and implementation of oral care calendar Patients in the intervention group were given a calendar for documenting their oral care practices. With this calendar, the child and their caregiver and the nurse had the opportunity to track oral care practices.

Figure 4. Followed Oral Care Calendar and Training Children in the intervention group who applied and completed the care protocol for 14 days received a certificate of appreciation prepared by the researchers

Stage 4: Implementation of oral care protocol Within the scope of the study, the oral care protocol prepared on the basis of the literature was applied to the intervention group over a 14-day period. Laboratory values were monitored, and the application was evaluated during the application process.

Prior to treatment (Day 0), each child in the intervention group underwent an oral examination. Following the results of the evaluation, participants were instructed to gargle with sodium bicarbonate (5 cc) six times per day starting on Day 1 and to gargle and spit between meals. They received mouthwash with sodium chloride (5 cc) to be spit and Mycostatin (2 cc) to be swallowed after each meal. They were also asked to gargle and swallow glutamine (5 cc) three times a day before or between meals. Together with the caregiver, each participant was instructed to use dental floss after eating twice per day and then brush their teeth with a soft toothbrush and fluoride toothpaste. The American Academy of Pediatric Dentistry recommends brushing the teeth unless bleeding occurs. The American Academy of Pediatric Dentistry (2022) advises patients to maintain good oral hygiene by brushing their teeth and tongue two to three times a day, regardless of their hematological status. Flossing is reportedly effective in preventing oral mucositis but should be done under the guidance of a caregiver (Ferrández-Pujante, 2022). Finally, the participants were told to use Lanolin-containing lip moisturizer at least twice a day and to not eat or drink for half an hour after applying the moisturizer. Table 1 presents the daily oral care practice for the intervention group. Evaluations were performed on Days 0, 3, 7, and 14 of the application.

Control Group Children in the control group will receive standard care. Mouthwash with sodium bicarbonate (after each feeding), mycostatin (2x1) and tranflex (3x1). Toothbrush and dental floss are not used. At the end of the 14th day, the child and caregiver in the control group will receive Oral Care Protocol Training to Prevent Oral Mucositis.

ELIGIBILITY:
Inclusion criteria:

* Being between 6 and 18 years,
* Having received at least 1 course of chemotherapy,
* Having no visual, auditory, or intellectual problems
* Speaking and understanding Turkish
* Being willing to participate in the research.

Exclusion criteria:

-Conditions that prevent verbal communication (neurodevelopmental delay, verbal speech difficulties, hearing or hearing problems; oral mucositis).

Ages: 6 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
CHIMES scores | day0
  The scale consists of categories such as the severity of pain in the mouth, the effect of pain on swallowing, eating, drinking, taking painkillers, and the presence of ulcers in the mouth.The lowest score obtained from the scale is 0, the highest score is 23. The higher the total score, the more advanced the degree of mucositis
CHIMES scores | day3
  The scale consists of categories such as the severity of pain in the mouth, the effect of pain on swallowing, eating, drinking, taking painkillers, and the presence of ulcers in the mouth.The lowest score obtained from the scale is 0, the highest score is 23. The higher the total score, the more advanced the degree of mucositis
CHIMES scores | day7
  The scale consists of categories such as the severity of pain in the mouth, the effect of pain on swallowing, eating, drinking, taking painkillers, and the presence of ulcers in the mouth.The lowest score obtained from the scale is 0, the highest score is 23. The higher the total score, the more advanced the degree of mucositis
CHIMES scores | day14
  The scale consists of categories such as the severity of pain in the mouth, the effect of pain on swallowing, eating, drinking, taking painkillers, and the presence of ulcers in the mouth.The lowest score obtained from the scale is 0, the highest score is 23. The higher the total score, the more advanced the degree of mucositis
WHO Oral Mucositis Granding Scale | day0
  The presence of oral mucositis is assessed based on clinical manifestations. The score ranges from 0 (the absence of manifestations and symptoms) to 4 (oral feeding is impossible). Grade-0 no change in mucosa, Grade-1 painless ulcers, erythema or mild sensitization, Grade-2 painful erythema and ulcer but can consume solid foods. Grade-3 painful erythema, edema or ulcer can consume only fluids, Grade-4 ulceration, necrosis and hemorrhage, patient cannot feed, enteral or parenteral support is required
WHO Oral Mucositis Granding Scale | day3
  The presence of oral mucositis is assessed based on clinical manifestations. The score ranges from 0 (the absence of manifestations and symptoms) to 4 (oral feeding is impossible). Grade-0 no change in mucosa, Grade-1 painless ulcers, erythema or mild sensitization, Grade-2 painful erythema and ulcer but can consume solid foods. Grade-3 painful erythema, edema or ulcer can consume only fluids, Grade-4 ulceration, necrosis and hemorrhage, patient cannot feed, enteral or parenteral support is required
WHO Oral Mucositis Granding Scale | day7
  The presence of oral mucositis is assessed based on clinical manifestations. The score ranges from 0 (the absence of manifestations and symptoms) to 4 (oral feeding is impossible). Grade-0 no change in mucosa, Grade-1 painless ulcers, erythema or mild sensitization, Grade-2 painful erythema and ulcer but can consume solid foods. Grade-3 painful erythema, edema or ulcer can consume only fluids, Grade-4 ulceration, necrosis and hemorrhage, patient cannot feed, enteral or parenteral support is required
WHO Oral Mucositis Granding Scale | day14
  The presence of oral mucositis is assessed based on clinical manifestations. The score ranges from 0 (the absence of manifestations and symptoms) to 4 (oral feeding is impossible). Grade-0 no change in mucosa, Grade-1 painless ulcers, erythema or mild sensitization, Grade-2 painful erythema and ulcer but can consume solid foods. Grade-3 painful erythema, edema or ulcer can consume only fluids, Grade-4 ulceration, necrosis and hemorrhage, patient cannot feed, enteral or parenteral support is required

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Training and Research Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the participants are children, they are not wanted to share.